CLINICAL TRIAL: NCT05168228
Title: Evaluating the Long-term Neurocognitive Effects of Preconceptional Exposure to Iodinated Contrast During Hysterosalpingography (HSG) on the Offspring of the H2Oil Trial
Brief Title: Evaluating the Long-term Neurocognitive Effects of Preconceptional Exposure to Iodinated Contrast on the Offspring
Acronym: Neuro-H2Oil
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Velja Mijatovic, Professor in Obstetrics and Gynaecology, Specialist in Reproductive Medicine, Head of Endometriosis Center VUmc, Amsterdam UMC, location VUmc
Other Study IDs: 2021.0448
Record Dates: First submitted 2021-11-25; First posted 2021-12-23 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Neurocognitive Disorders
Keywords: Hysterosalpingography; Iodinated contrast media; Iodine; Intelligence; Neurocognitive development
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Oil- versus waterbased contrast in hysterosalpingography (HSG) — The Neuro-H2Oil study looks at the offspring of the H2Oil study, a randomized controlled trial (RCT) comparing hysterosalpingography (HSG) with oil- versus water-based contrast during fertility work-up. For more information please see NTR 3270 (original H2Oil study), www.trialregister.nl. The control group is the Database for Controls in Neuroscience Studies (D-CNS), registered as NL9574 (https://www.trialregister.nl/trial/9574).

SUMMARY:
Iodinated contrast is commonly used in hysterosalpingography (HSG), a diagnostic tool in fertility work-up. This study aims to investigate the safety of contrast media used during HSG by evaluating the long-term effects on the neurodevelopment of offspring 6-8 years after exposure to iodinated contrast media.

DETAILED DESCRIPTION:
Background: Iodinated contrast is commonly used in hysterosalpingography (HSG), a diagnostic tool in fertility work-up. Yet excessive iodine may pool for a long time in the body, crosses the placenta easily, and can induce hypothyroidism in both mothers and foetuses. Inadequate supplies of thyroid hormones have previously been associated with neurocognitive impairments in offspring. Considering the widespread use of iodinated contrast during fertility work-up, the potential iatrogenic effect of preconceptional iodine exposure on the brain development of the offspring needs to be addressed urgently.

Objectives: This project aims to investigate the safety of contrast media used during HSG by evaluating the long-term effects on the neurodevelopment of offspring 6-8 years after exposure to iodinated contrast media. To do this, the investigators will follow up on a cohort of offspring conceived during the H2Oil randomised controlled trial (NTR 3270), which was set up to evaluate the effect of using water- or oil-based media during HSG on pregnancy rates.

Methods: The study team have previously obtained parental permission for follow-up research in 140 children conceived during the H2Oil study <6 months after exposure to iodine during the HSG. The investigators will conduct comprehensive an in-depth outcome assessment of intelligence, neurocognitive development, school performance, and behavioural functioning.

Relevance: Using this diverse range of methods, the investigators expect to be the first to shed light on the long-term iatrogenic consequences of using iodinated contrast just before conception on the neurodevelopment of their offspring. The findings of this study will have implications for current clinical practice, where HSG is readily used in subfertile women, and will be used to inform the Dutch guidelines for fertility work-up.

ELIGIBILITY:
Inclusion Criteria:

* Children conceived after the mother underwent HSG procedure in the context of the H2Oil trial (2012-2014)
* Children must be conceived <6 months after the HSG procedure
* Parents must have given consent for recontacting for follow up research

Exclusion Criteria:

* Children conceived after the mother underwent HSG procedure that was not part of the H2Oil trial
* Children conceived >6 months after the HSG procedure
* Children whose parents did not give permission to be recontacted for follow up research
* Children that are not able to comprehend the instructions at the time of assessment
* Absence or withdrawal of written informed consent
* Inability to comprehend testing instructions at time of assessment
* Severe motor disability that interferes with outcome assessment at time of assessment
* Documented and/or parent-reported diagnosis of a neurological disorder
* Somatic disorders known to affect the outcome assessments at time of assessment

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children born to mothers who participated in the original H2Oil study (NTR3270), a multicentre randomised controlled trial on oil- versus water-based HSG in 2012-2014 whose parents gave consent to be contacted for follow up studies (n=140).
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
School performance | Between the ages of 4-12, up to 12 years
  Longitudinal data on school performance will be collected using standardised tests from the pupil monitoring system developed by the Dutch National Institute for Educational Measurement (CITO-test). CITO-tests are used to assess children's academic performance (reading comprehension, spelling, and arithmetic performance) in primary schools in the Netherlands.
Intelligence | 1 Day
  General intelligence will be assessed using a shortened Fifth version of the Wechsler Intelligence Scale for Children. Full-scale IQ (FSIQ) will be estimated using the subtests Vocabulary, Similarities, Matrix Reasoning, and Block Design.
Behavioural functioning evaluated through the Strengths and Difficulties Questionnaire (SDQ). | 1 Day
  Behavioural functioning will be evaluated through the Strengths and Difficulties Questionnaire (SDQ). Both parents and teachers will fill in the SDQ.
Behavioural functioning evaluated through the Strengths and Weaknesses of ADHD Symptoms And Normal behaviour (SWAN) scale. | 1 Day
  Behavioural functioning will be evaluated will be evaluated using the Strengths and Weaknesses of ADHD Symptoms And Normal behaviour (SWAN) scale. Both parents and teachers will fill in the SWAN scale.

SECONDARY OUTCOMES:
Visuomotor integration | 1 Day
  Visuomotor integration will be assessed using a Track & Trace task of the Emma Toolbox for Neurocognitive Functioning, which is an in-house designed battery of computerised tests for assessing different neurocognitive domains.
Processing & Control | 1 Day
  Processing & Control will be assessed using an Attention Network Test of the Emma Toolbox for Neurocognitive Functioning, which is an in-house designed battery of computerised tests for assessing different neurocognitive domains.
Visual Memory | 1 Day
  Visual Memory will be assessed using an Location Learning Test of the Emma Toolbox for Neurocognitive Functioning, which is an in-house designed battery of computerised tests for assessing different neurocognitive domains.
Verbal Memory | 1 Day
  Verbal Memory will be assessed using a Rey Auditory Verbal Learning Test (Dutch Version) of the Emma Toolbox for Neurocognitive Functioning, which is an in-house designed battery of computerised tests for assessing different neurocognitive domains.
Visual Working Memory | 1 Day
  Visual Working Memory will be assessed using a Klinberg task of the Emma Toolbox for Neurocognitive Functioning, which is an in-house designed battery of computerised tests for assessing different neurocognitive domains.
Verbal Working Memory | 1 Day
  Verbal Working Memory will be assessed using a Digit Span task of the Emma Toolbox for Neurocognitive Functioning, which is an in-house designed battery of computerised tests for assessing different neurocognitive domains.

CONTACTS AND LOCATIONS:
Overall Officials: Marsh Königs, PhD, Principal Investigator — Emma Children's Hospital, Amsterdam UMC
Locations (1):
- Emma Kinderziekenhuis, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Konigs M, Verhoog EM, Oosterlaan J. Exploring the neurocognome: Neurocognitive network organization in healthy young adults. Cortex. 2021 Oct;143:12-28. doi: 10.1016/j.cortex.2021.06.011. Epub 2021 Jul 14. PMID 34365200
- [Background] Dreyer K, van Rijswijk J, Mijatovic V, Goddijn M, Verhoeve HR, van Rooij IAJ, Hoek A, Bourdrez P, Nap AW, Rijnsaardt-Lukassen HGM, Timmerman CCM, Kaplan M, Hooker AB, Gijsen AP, van Golde R, van Heteren CF, Sluijmer AV, de Bruin JP, Smeenk JMJ, de Boer JAM, Scheenjes E, Duijn AEJ, Mozes A, Pelinck MJ, Traas MAF, van Hooff MHA, van Unnik GA, de Koning CH, van Geloven N, Twisk JWR, Hompes PGA, Mol BWJ. Oil-Based or Water-Based Contrast for Hysterosalpingography in Infertile Women. N Engl J Med. 2017 May 25;376(21):2043-2052. doi: 10.1056/NEJMoa1612337. Epub 2017 May 18. PMID 28520519
- [Derived] Keestra SM, Van Welie N, Dreyer K, Van Eekelen R, Roseboom TJ, Oosterlaan J, Mol BW, Finken MJJ, Mijatovic V, Konigs M. Neurodevelopmental outcomes of school-age children conceived after hysterosalpingography with oil-based or water-based iodinated contrast: long-term follow-up of a nationwide randomized controlled trial. Hum Reprod. 2024 Oct 1;39(10):2287-2296. doi: 10.1093/humrep/deae183. PMID 39198011